CLINICAL TRIAL: NCT06269211
Title: Neoadjuvant Toripalimab for Clinically Stage II-IIIB Resectable Non-small Cell Lung Cancer with EGFR Mutation and PD-L1 Positive Expression: a Prospective, Open-label, Multicenter, Single-arm Phase II Clinical Study
Brief Title: Neoadjuvant Toripalimab for Clinically Stage II-IIIB Resectable Non-small Cell Lung Cancer with EGFR Mutation and PD-L1 Positive Expression
Acronym: TOPLINE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Chair of thoracic department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-019
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: This study has only one arm, neoadjuvant Toripalimab treatment arm. Primary endpoint is MPR. We apply the optimal design of Simon's two-stage model to calculate the sample size and set both sides α= 0.05 and power=0.8, resulting in a total sample size of 29. Among them, 10 patients will be enrolled in the first stage. If the number of MPR cases in the first stage is less than or equal to 1, the study will be terminated in the early stage; On the contrary, participants in the second stage will continue to be enrolled. If the total number of MPR cases is greater than or equal to 5 after the completion of the second stage, the study is considered positive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab (Experimental): Neoadjuvant Toripalimab 240 mg IV on cycle 1 day 1 (C1D1), C2D1 and C3D1 before radical surgery for lung cancer. The participants will attend follow-up visits based on molecular residual disease (MRD) and receive adjuvant treatment including EGFR-TKI or chemotherapy if recommended.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — 240mg IV, Q3W

SUMMARY:
The study is a prospective, open label, multicenter, single arm Phase II clinical trial, aiming to explore the use of neoadjuvant Toripalimab for clinically stage II-IIIB NSCLC patients with EGFR mutations and PD-L1 positive expression, providing a novel perspective for further improving the prognosis of NSCLC patients. This study will provide valuable information for further clinical trials of neoadjuvant Toripalimab and other immune checkpoint inhibitors in NSCLC patients with EGFR mutations and PD-L1 positive expression.

DETAILED DESCRIPTION:
For resectable locally advanced non-small cell lung cancer (NSCLC), the combination of neoadjuvant therapy and surgery has benefited the patients and has become a clinical routine and guideline recommended treatment. Among the East Asian NSCLC population, about 30% are positive for EGFR driver gene mutations. The efficacy of this population receiving neoadjuvant chemotherapy and EGFR inhibitors is limited, and their optimal neoadjuvant treatment strategy is still unclear. The neoadjuvant immunotherapy has achieved good therapeutic effects in driver-negative NSCLC patients, and is superior in PD-L1 expression positive patients.

Based on the above evidence, the investigators plan to conduct a prospective, open label, multicenter, single arm Phase II clinical study to explore the use of neoadjuvant Toripalimab for clinically stage II-IIIB NSCLC patients with EGFR mutations and PD-L1 positive expression, providing a novel perspective for further improving the prognosis of NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥ 18 years old.
2. Baseline tumor tissues have to be obtained through biopsy (percutaneous or transbronchial) or surgery at study center.
3. Histologically confirmed diagnosis of primary non-small lung cancer on non-squamous histology.
4. Pre-treatment stage as clinical II-IIIB (AJCC/UICC 8th Edition) (stage IIIB excludes N3 disease); curative resectability has to be explicitly verified by the experienced surgical investigator.
5. Confirmation by the central laboratory that the tumor harbors EGFR mutations either sensitive mutations, uncommon mutations or complex mutations.
6. Have a PD-L1 tumor proportion score (TPS) ≥ 1% determined by IHC at the central laboratory. In order to balance patients with high PD-L1 expression (≥50%) and low PD-L1 expression (1-49%), we planned to enroll PD-L1 high and low patients at a ratio of 1:1.
7. Have not received prior systemic treatment for NSCLC.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
9. Expected survival ≥ 3 months.
10. Adequate blood and organ function.

Exclusion Criteria:

1. Patients with histologically confirmed squamous cell carcinoma, combined small cell carcinoma and large cell carcinoma.
2. Molecular testing confirmed ALK translocation.
3. Treatment with prior systemic cancer therapy for the current lung cancer at any time (chemotherapy, radiotherapy, target therapy, ablation, and any other local or systemic therapy).
4. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colorectal, endometrial, cervical, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
5. Any active or history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications. Subjects with vitiligo, type I diabetes mellitus, resolved childhood asthma/atopy, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement or unexpected conditions of recurrence in the absence of an external trigger are allowed to be included.
6. Subjects with a history of interstitial lung disease, pneumonitis, or poorly controlled lung disease (including pulmonary fibrosis, acute lung diseases).
7. Severe chronic or active infections that require systemic antimicrobial, antifungal, or antiviral treatment, including tuberculosis infections.
8. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA ≥ 500 IU/mL [2500 copies/mL] should be excluded.
9. Has known active hepatitis C virus (HCV). Active HCV is defined by positive tests for HCV Ab and quantitative HCV RNA.
10. Known positive history or positive test for Human Immunodeficiency Virus (HIV).
11. The investigator believes that there is a high risk of bleeding (such as esophageal varices with bleeding risk, local active ulcer lesions) or active hemoptysis.
12. History of allergy to study drug components.
13. Pregnant and lactating women are excluded.
14. Fertile men or their female partners (women of childbearing potential, WOCBP) who are not willing to use contraception.
15. Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information.
16. The investigator believes that there are factors that can increase medication risk or confuse outcome judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | MPR will be assessed within 2 weeks after surgery
  Defined as the incidence rate in postoperative pathology where the percentage of surviving tumor cells in the tumor bed is ≤ 10%, regardless of the presence or absence of live tumor cells in the lymph nodes.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | pCR will be assessed within 2 weeks after surgery
  Defined as the proportion of patients in postoperative pathology who have no residual live tumor cells in the primary tumor bed or in all excised lymph nodes.
Objective Response Rate (ORR) | Tumor response will be evaluated within 30 days after last dose of neoadjuvant treatment
  Based on the solid tumor evaluation criteria (RECIST 1.1), the sum of the proportions of complete and partial remission evaluated by imaging
2-year Event Free Survival (EFS) | 2 years after the date of initiation of neoadjuvant treatment
  EFS is defined as the time from the first use of the investigational drug to any of the following events (whichever occurs first): the investigator assessed the disease progression based on imaging according to RECIST 1.1 and therefore was unable to receive curative surgery, local or distant recurrence, or death from any cause. A 2-year EFS is used as a secondary endpoint.
2-year Overall Survival (OS) | 2 years after the date of initiation of neoadjuvant treatment
  OS is defined as the date from the first use of the investigational drug until death from any cause. A 2-year OS is used as a secondary endpoint.
Safety (Number of Participants With Grade 3 and Higher-grade Treatment-related Adverse Events) | From date of neoadjuvant treatment until surgery was applied during study period or up to at least 90 days after last dose.
  The safety evaluation will be based on weekly blood routine tests, liver and kidney function, electrolyte analysis, etc., and adverse reactions of level 3 or above will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE 5.0).
Feasibility (Number of Participants Who Finished Neoadjuvant therapy and Receive Surgery Within 3-6 Weeks After Neoadjuvant Therapies) | 6 weeks after last dose of neoadjuvant treatment
  Among patients who have been evaluated as operable after completing neoadjuvant therapy, a surgical period of no more than 42 days from the completion of neoadjuvant therapy is defined as feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, PhD, MD, Principal Investigator — Ruijin hospitalRuijin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No